CLINICAL TRIAL: NCT00242359
Title: A Pilot Study Investigating the Effect of Omalizumab (Xolair) in Work-Related Animal Induced Asthma
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: could not find subject population
Sponsor: Bernstein Clinical Research Center (Other)
Responsible Party: Principal Investigator, Jonathan A. Bernstein, MD, principal investigator, Bernstein Clinical Research Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2085
Record Dates: First submitted 2005-10-17; First posted 2005-10-20 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Allergy Induced Asthma
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- omalizumab (Other): open-label
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab

SUMMARY:
Management of animal induced occupational asthma is mainly avoidance, but this is not feasible for many occupations. Treatment with avoidance and conventional treatment is also not always successful. Omalizumab is FDA approved for the treatment of allergic asthma and may be effective at reducing symptoms and disease progression in the animal handlers population.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-65
2. occupation that involves close contact with animals
3. stable dose of ICS for 30 days
4. Skin test positive to one or more animals
5. evidence of asthma on spirometry
6. demonstrate PEFR variability-

Exclusion Criteria:

1. on allergen immunotherapy
2. on prohibited medications
3. unstable asthma
4. recent URI
5. known hypersensitivity to omalizumab-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)